CLINICAL TRIAL: NCT06839352
Title: Assessment of Efficacy and Safety of Intravenous Vitamin K1 in Management of Acute Variceal Bleeding in Patients With Liver Cirrhosis: A Randomized Open Label Clinical Trial
Brief Title: Efficacy and Safety of Intravenous Vitamin K1 in Management of Acute Variceal Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ayman Magd Eldin Mohammad Sadek, Associate Professor of Internal Medicine, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#9092/16-11-2021
Record Dates: First submitted 2025-01-27; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Variceal Bleeding
Keywords: Vitamin K1; Liver cirrhosis; Esophageal and gastric varices; Upper gastrointestinal bleeding
MeSH Terms: conditions — Liver Cirrhosis; Esophageal and Gastric Varices; Gastrointestinal Hemorrhage | interventions — Vitamin K 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin K1 (Active Comparator)
  Interventions: Drug: Vitamin K1
- Control (No Intervention)

INTERVENTIONS:
Drug: Vitamin K1 — 10 mg intravenous infusion daily for three days
  Arms: Vitamin K1

SUMMARY:
The administration of Vitamin K1 (Vit-K1) injection is frequently utilized in clinical practice for managing upper gastrointestinal bleeding (UGIB) associated with liver cirrhosis, despite insufficient evidence supporting its effectiveness. This research aimed to assess the safety and efficacy of intravenous Vit-K1 in the management of acute variceal bleeding in cirrhotic patients.

This randomized, open-label clinical trial involved 66 cirrhotic cases with UGIB of suspected variceal origin. The cases were randomly assigned to two groups: one group (n = 33) had a 10 mg intravenous infusion of Vit-K1 daily for three days, while the other group (n = 33) received nothing, along with standard pharmacologic and endoscopic treatments. Endoscopic evaluation confirmed ruptured varices as the cause of bleeding in 59 cases. The primary endpoint was a composite measure that involved (bleeding control, rebleeding prevention, or death).

Adding vitamin K1 to standard-of-care therapy in managing acute variceal bleeding complicating liver cirrhosis showed no advantage over standard-of-care therapy in terms of bleeding control, prevention of rebleeding, or reducing mortality during hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Active acute upper gastrointestinal bleeding suspected of being of variceal origin (e.g., melena and/or hematemesis within 24 hours before inclusion) and required admission to the ICU.
* Endoscopic confirmation of variceal bleeding, carried out within twelve to twenty-four hours of ICU admission, was defined by either direct visualization of blood from a gastric or esophageal varix or the presence of red color signs on varices along with blood in the stomach or esophagus, with no other identifiable bleeding source.
* Cirrhosis has been confirmed through histology or by clear clinical, endoscopic, or sonographic signs of portal hypertension and cirrhosis.

Exclusion Criteria:

* Known hypersensitivity to Vit-K1.
* Known hypercoagulopathy.
* Recent history (within 6 months) including deep vein thrombosis or pulmonary embolism.
* History of persistent or unstable angina pectoris, portal vein thrombosis, intermittent claudication, myocardial infarction, ischemic stroke, transient ischemic attack.
* Prior parenteral or oral Vit-K1 administration within the previous two weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Number of patients failed to control bleeding | 1st 6 hours - from 6 to 24hours - from 24 hours to 5 days
Number of patients with rebleeding | within 5 days
Number and percent of mortality | 5 days

SECONDARY OUTCOMES:
Median (IQR) of length of ICU staying | 7 days
Median (IQR) of length of hospital stay | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Sadek, MD, Study Chair — Zagazig University
Locations (1):
- Zagazig University Hospital, Zagazig, Sharqia Province, Egypt